CLINICAL TRIAL: NCT06363110
Title: Titration Patterns, Patient Characteristics and Hypotension Events Among Patients Initiating Vericiguat in Real World Settings in the United States (US)
Brief Title: An Observational Study to Learn More About Vericiguat Treatment Patterns and Its Safety in People With Chronic Heart Failure With Reduced Ejection Fraction in Routine Medical Care in the United States
Acronym: HOVER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22724
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients initiating vericiguat: Adult patients initiating vericiguat in the US. Retrospective single-arm cohort analysis using HealthVerity Heart Failure (HF) dataset licensed by Bayer.
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — Follow clinical practice/administration

SUMMARY:
This is an observational study in which data already collected from people with chronic heart failure with reduced ejection fraction (HFrEF) are studied.

In observational studies, only observations are made, without participants receiving any advice or any changes to healthcare.

Chronic HFrEF is a long-term condition in which the heart becomes weak and cannot pump enough blood to the rest of the body with each heartbeat. This leads to a reduced supply of oxygen, which the body requires to function properly.

The study treatment, vericiguat, works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC), which relaxes the blood vessels and allows more blood to flow. As a result, the heart can pump better.

It is already approved for doctors to prescribe to people with chronic HFrEF in the United States (US) who are stabilized after a recent "decompensation event". The treatment with vericiguat starts at a low dose, which should be increased gradually to the target dose based on how a patient tolerates the treatment.

The participants in this study are already receiving treatment with vericiguat as part of their regular care from their doctors.

The main purpose of the study is to learn more about the dosage pattern of vericiguat in people with chronic HFrEF in the US. To do this, researchers will collect the following information for 3 months after participants' first dose of vericiguat:

* starting dose of vericiguat
* daily changes in dosage pattern
* time taken to reach the target dose
* number and percentage of participants:
* with specific changes in dosage pattern
* reaching the target dose of vericiguat

They will also collect information on how often low blood pressure or fainting occurs, which are well known events in people with chronic HFrEF.

The data will come from the participants' information stored in a database called the HealthVerity HF dataset. Data collected will be from people with chronic HFrEF who started taking vericiguat between January 2021 and April 2023.

Researchers will only look at the health records of participants in the US.

Researchers will track participants' data and will collect information for a maximum of 6 months before and 3 months after their first dose of vericiguat.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first vericiguat fill from a closed pharmacy claim, defined as the index date, during the patient identification period spanning from 01 JAN 2021 - 01 APR 2023.
* Patients aged 18 years or older at index date.
* Patients with at least 180 days of medical and pharmacy enrollment (no gap) prior to index date (inclusive).

Exclusion Criteria:

* Patients with any open pharmacy claim in the 180-day prior to index date
* Patients with an open pharmacy claim for vericiguat at index date and in the 90 days after index date
* Patients with missing age (last value observed) and gender (last value observed) at index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who initiated vericiguat from closed claims during 01Jan2021 and 01Apr2023 and who have at least 6 months of prior observability.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Number of patients having vericiguat daily dose of 2.5 mg, 5 mg and 10 mg at index date | Retrospective data analysis from 01Jan2021 to 01Apr2023
Number of patients having daily dose of 10 mg/day within the 90 days after vericiguat initiation | Retrospective data analysis from 01Jan2021 to 01Jul2023
Days from index date to first occurrence of 10 mg/day dose | Retrospective data analysis from 01Jan2021 to 01Jul2023
Number of patients who received a dose of 2.5 mg/day, 5 mg/day and 10 mg/day, or discontinued drug therapy each day over the 90-day follow-up period | Retrospective data analysis from 01Jan2021 to 01Jul2023
Number of patients having any Vericiguat up-titration within the 90 days after vericiguat initiation | Retrospective data analysis from 01Jan2021 to 01Jul2023
  Vericiguat up-titration is defined as first vericiguat prescription with a higher dose compared to the previous vericiguat prescription:
  * 2.5 mg/day at index date followed by any dose >2.5 mg/day during follow-up, OR
  * 5 mg/day at index date followed by any dose >5 mg/day during follow-up
Number of patients having specific titration scenarios within the 90 days after vericiguat initiation | Retrospective data analysis from 01Jan2021 to 01Jul2023
  7 titration patterns:
  * Vericiguat dose of 2.5 mg/day at index date, without 5 mg/day dose and without 10 mg/day dose observed during follow-up
  * Vericiguat dose of 2.5 mg/day at index date followed by 5.0 mg/day dose during follow-up and without 10 mg/day dose observed during follow-up
  * Vericiguat dose of 2.5 mg/day at index date, followed by 5 mg/day dose, and followed by 10 mg/day dose during follow-up
  * Vericiguat dose of 5.0 mg/day at index date without 10 mg/day dose observed during follow-up
  * Vericiguat dose of 5 mg/day at index date followed by 10 mg/day dose during follow-up
  * Vericiguat dose of 2.5 mg/day at index date, followed by 10 mg/day dose and without 5 mg/day dose observed during follow-up
  * Vericiguat dose of 10 mg/day at index date without 2.5 mg/day dose and without 5 mg/day dose observed during follow-up

SECONDARY OUTCOMES:
Number of patients having hypotension or syncope in the entire 90 days after vericiguat initiation and by 30 days intervals | Retrospective data analysis from 01Jan2021 to 01Jul2023

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.